CLINICAL TRIAL: NCT06857929
Title: Nutritional Approach for the Transformation and Reduction of Chronic Disease Indicators in Middle-aged Adults at High Risk
Brief Title: "Improving Health and Reducing Chronic Disease Risk in Middle-Aged Adults Through Nutrition"
Acronym: NUTRI-M-Care
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: IMDEA Food (Other)
Responsible Party: Principal Investigator, Lidia Daimiel Ruiz, Principal Investigator, IMDEA Food
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IMD PI-071
Record Dates: First submitted 2025-03-03; First posted 2025-03-05 (Actual); Last update posted 2025-04-25 (Actual); Status verified 2025-04

CONDITIONS: Metabolic Syndrome; Obesity Prevention; Obesity and Overweight
Keywords: metabolic syndrome; Mediterranean diet; Caloric restriction; Physical activity; Weight loss; Weight; body composition
MeSH Terms: conditions — Metabolic Syndrome; Obesity; Overweight; Motor Activity; Weight Loss; Body Weight | interventions — Caloric Restriction; Exercise

STUDY DESIGN:
Intervention Model Description: It is a randomized, controlled, single blinded, parallel group clinical trial aiming to evaluate the effect of a multifactorial intervention based on Mediterranean diet, energy reduction and physical activity on parameters of metabolic syndrome in middle-aged men and women.
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control group (CG) (Active Comparator): The aim of this group is to serve as control comparator of the intervention. Participants allocated to this group will be asked to follow genera lifestyle recommendations included in the clinical guidelines for metabolic syndrome in primary healthcare settings
  Interventions: Behavioral: Usual Care
- Intervention Group (IG) (Experimental): Participants in this group will be asked to follow an energy-reduced Mediterranean diet and a physical activity program with the aim of lossing 5-10% of the initial weight in 6 months
  Interventions: Behavioral: energy reduced Mediterranean diet (25% caloric restriction) plus physical activity program

INTERVENTIONS:
Behavioral: energy reduced Mediterranean diet (25% caloric restriction) plus physical activity program — An intensive multifactorial lifestyle intervention involving monthly individual and group sessions during 6 months. Participants will be asked to follow a Mediterranean diet with a 25% reduction in energy and a physical activity program based on WHO recommendations to achieve a moderate physical activity level.
  Other Names: Multifactorial lifestyle intervention; energy-reduced mediterranean diet; Physical activity; Caloric restriction
  Arms: Intervention Group (IG)
Behavioral: Usual Care — Participants in the control group will be asked to follow general recommendations to adhere to a healthy lifestyle, as indicated in the clinical guidelines of general practitioners and nurses for adults with metabolic syndrome
  Arms: Control group (CG)

SUMMARY:
The goal of this clinical trial is to evaluate the effect of a multifactorial lifestyle intervention combining Mediterranean diet, energy reduction and physical activity on weight loss in middle-aged adults (men and women 30-50 years old) with metabolic syndrome. The main questions it aims to answer are:

Is a multifactorial intervention based on Mediterranean diet, energy reduction and physical activity able to promote weight loss maintenance in middle-aged men and women with metabolic syndrome? syndrome? Which are the sociodemographic barriers to adhere to a multifactorial lifestyle intervention to promote cardiometabolic health? How is the lifestyle pattern of middle-aged Spanish adults with metabolic

Researchers will compare a multifactorial lifestyle intervention combining Mediterranean diet, energy reduction and physical activity to a control intervention based on usual primary healthcare to see if the intervention improve cardiometabolic traits and promote weight loss maintenance after 1 year.

Participants in the intervention arm will be asked to follow an energy-reduced Mediterranean diet plus a physical activity program with the aim of reducing 5-10% of the initial weight in 6 months and of maintaining the weight lost after 1 year o follow-up.

DETAILED DESCRIPTION:
Metabolic syndrome (MetS), characterized by the presence of hyperglycemia, hypertension, abdominal obesity and dyslipidemia, is associated with the development of non-communicable diseases such as cardiovascular disease, diabetes or different types of cancer. The prevalence of MetS is increasing in the population. Most of the affected population is elderly adult population (> 50 years), although the incidence of MetS in young adults is growing at a worrying rate. The presence of MetS is associated with chronic medication and has a great impact on the quality of life of individuals, but it also has a huge socioeconomic impact on the population. Therefore, implementing strategies aimed at preventing MetS at an early age is of crucial importance for maintaining population health.

Adopting healthier lifestyle habits has been shown to be a protective measure against MetS. Pursuing these changes to become part of people's daily routines takes time and they always face various obstacles along the way. There are 4 phases before achieving this change: one of mind reflection, another of preparation, one of action and finally maintenance.

The present study attempts, with middle-aged adult patients with MetS, to influence these 4 phases and evaluate whether changes in eating habits, more specifically, adherence to a Mediterranean diet with energy restriction, and physical activity, promoted within the frame of Primary Care have an impact on the reversal and control of such pathology: on the one hand, whether the general well- being of the participants is improved and how positive the changes are in the metabolic, anthropometric, analytical and cardiovascular health parameters and, on the other hand, the effect that occurs on nutrient intake and the overall dietary pattern. Moreover, without neglecting the maintenance phase that seeks to identify facilitators and impediments for its long-term maintenance outside the spectrum of action of the study.

The study will be an open, controlled, randomized clinical trial with parallel groups, made up of adults between 30 and 50 years of age with MetS, with one group in intervention for 6 months and one control group with recommendations from nursing clinics for populations with chronic diseases and/or analytical disorders. In month 12, 6 months after the completion of the intervention for each patient in the study, an evaluation of adherence to the therapeutic plan will be carried out of the group independently.

Data collection during the trial will be of 3 types: sociodemographic, anthropometric, dietary, clinical and analytical. Our hypothesis is that a change in diet and physical activity, promoted from the area of Primary Care in the young adult population with MetS, impacts the following aspects: encourage reflection on the need to change lifestyle habits; prepare the patient to make modifications aimed at improving their well-being; guide on the actions necessary to achieve the reversal and management of MetS and maintain life changes once the study is completed.

ELIGIBILITY:
Inclusion Criteria:

* BMI 27-40 Kg/m2
* Metabolic syndrome according to International Diabetes Federation Task Force on Epidemiology and Prevention; National Heart, Lung, and Blood Institute; American Heart Association; World Heart Federation; International Atherosclerosis Society; and International Association for the Study of Obesity
* Stable weight in the last 3 months (weight changes < 4Kg)
* Be able to give informed consent

Exclusion Criteria:

* Have a diagnosed illness that interferes with the recommendations proposed in the intervention.
* Women with established menopause.
* Pregnant or breastfeeding women.
* Serious psychiatric illness/disorder.
* Social, cultural or psychological factors that may affect adherence to the intervention protocol.
* Inability to communicate with study staff.
* Inability to follow recommended diet or inability to engage in physical activity.
* Low likelihood of modifying dietary habits according to the different stages of change according to the Prochaska and DiClemente model.
* Difficulty attending scheduled appointments within the intervention due to work schedule conflicts, travel plans, scheduled surgeries, among other reasons.
* Therapeutic non-compliance.
* Participating in a professionally-led nutritional intervention.
* Being under medical treatment that affects weight, intake or energy expenditure in the 3 months preceding the start of the study.

Smokers who have changed their smoking habit in the 6 months preceding the start of the study (including starting or stopping smoking).

- Participation in another trial that may interfere with this proposed study.

Ages: 30 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 106 (Estimated)
Dates: Start 2025-05-01 (Estimated); Primary Completion 2027-03-31 (Estimated); Study Completion 2028-08-31 (Estimated)

PRIMARY OUTCOMES:
Percentage of weight loss | 6 months
  Weight loss measured as % from baseline weight with a calibrated scale
Percentage of weight loss maintenance | 12 months
  Percentage of weight loss maintained after 1 year, measured by a calibrated scale

SECONDARY OUTCOMES:
Change in waist perimeter (cm) | 6 months
  Waist circumference change (cm) after 6 months, measured at the midpoint between the last rib and the iliac crest using a flexible tap
Changes in tryglyceride level | 6 months
  Changes in trlyglycerides (mg/dL) after 6 months, measured from an overnight fasting blood with standard analyticial methods
Changes in fasting glucose levels | 6 months
  Changes in glucose levels (mg/dL), measured from blood collected after an overnight fast using standard analytical methods
Changes in glycated hemoglobin | 6 months
  Changes in % of glycated hemoglobin, measured from blood collected after and overnight fast, by standard methods

CONTACTS AND LOCATIONS:
Overall Officials: Lidia Daimiel Ruiz, Senior Researcher, Principal Investigator — IMDEA Food

IPD SHARING:
Plan to Share IPD: Yes
All IPD data that underlie results in a publication may be shared with other researcher only for non-profit scientific purposes upon reasonable request.
  The study protocol and the statistical analysis plan will be made public through an official publication. The results of this clinical study will be published folowing Open-Science Principles.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: The protocol and the statistical analysis plan will be made publicly available at study recruitment ends. The IPD will be made accessible to other researcher 2 years after the publication of the main study outcomes
Access Criteria: Anonymised, coded data (sociodemographic, anthropometric, clinical and biochemical) may be accessible to other researchers only for non-profit scientific purposes and upon reasonable request to the principal investigator.